CLINICAL TRIAL: NCT00674115
Title: Randomized, Crossover Pharmacodynamic Study Comparing the Effects of Zegerid® (20 mg Omeprazole/Sodium Bicarbonate) and Prilosec OTC® (20 Mg-equivalent Omeprazole)
Brief Title: A Pharmacodynamic Study Comparing Zegerid® and Prilosec OTC® (CL2007-17 )(P07813)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 18133; CL2007-17; P07813 (Other: Merck)
Record Dates: First submitted 2008-05-02; First posted 2008-05-07 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-02

CONDITIONS: Gastric Acid; Human Experimentation
MeSH Terms: interventions — omeprazole, sodium bicarbonate drug combination; Omeprazole; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Dose Zegerid for 1 or 7 days (Experimental): Omeprazole 20 mg/Sodium Bicarbonate 1680 mg Powder for Oral Suspension
  Interventions: Drug: Omeprazole/sodium bicarbonate
- Single Dose Prilosec 1 or 7 days (Active Comparator): Omeprazole magnesium 20 mg over-the-counter (OTC) Tablet
  Interventions: Drug: omeprazole magnesium
- Sodium Bicarbonate (Active Comparator): Sodium Bicarbonate 1680 mg Oral Suspension
  Interventions: Drug: sodium bicarbonate

INTERVENTIONS:
Drug: Omeprazole/sodium bicarbonate — Omeprazole/sodium bicarbonate. Single dose per day for either 1 or 7 days.
  Other Names: Zegerid
  Arms: Single Dose Zegerid for 1 or 7 days
Drug: omeprazole magnesium — Omeprazole 20 mg tablet. Single dose per day for either 1 or 7 days.
  Other Names: Prilosec OTC Tablet
  Arms: Single Dose Prilosec 1 or 7 days
Drug: sodium bicarbonate — Sodium bicarbonate. Single dose.
  Arms: Sodium Bicarbonate

SUMMARY:
Open-label randomized crossover design studies. 60 participants will be evaluated on Day 1 to compare effects on stomach acid; 30 participants will continue treatment for 7 days and will have repeat evaluations at Day 7. The other 30 participants will receive a single administration of sodium bicarbonate.

DETAILED DESCRIPTION:
Enrolled participants were divided into 2 groups, with 30 participants in each group.

Group 1: This group was randomized into a 2-way crossover design with an added third period. These participants received single administrations (day 1 dosing only) of Zegerid Powder for Oral Suspension, and Prilosec OTC (both at a 20 mg omeprazole dose), in a 2-way randomized order, with a minimum of a 2-week washout period between treatment legs. Following completion of the 2-way crossover study, and a subsequent washout period (minimum of 2 weeks), all participants then received a single administration of sodium bicarbonate (at same dose as contained in Zegerid Powder for Oral Suspension) in Period 3. This group underwent a 24-hour intragastric pH study on each of the 3 dosing occasions.

Group 2: This group was randomized into a 2-way crossover design in which they received 7 days administration of Zegerid Powder for Oral Suspension and Prilosec OTC tablets, respectively. As with the prior group, there was a minimum of a 2-week washout period between treatment legs. Participants assigned to this treatment group also underwent 24-hour intragastric pH recordings on the days on which they received their 1st and last (7th) dose of the two treatment drugs.

In addition to the above detailed procedures, all participants (both groups) underwent a 24-hour baseline intragastric pH study prior to starting their randomized treatments. This study design enabled all 60 participants to be evaluated for effects of the first dose of Prilosec OTC and Zegerid Powder for Oral Suspension on change in intragastric pH during the subsequent 24-hour period following the first dose.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects who are 18-65 years of age.
* Non-childbearing potential females or those using birth control.

Exclusion Criteria:

* History of hypersensitivity, allergy or intolerance to omeprazole or other proton pump inhibitors
* History of significant gastrointestinal disease
* Any significant medical illness
* Gastrointestinal disorder or surgery leading to impaired drug absorption
* Currently using gastrointestinal medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 participants were randomized to either 1-Day or 7-Day Dosing in this crossover study (participants in both groups received 1 treatment [Zegerid or Prilosec], followed by washout period, followed by the other treatment [Prilosec or Zegerid]). Participants in the 1-day dosing group also received sodium bicarbonate after a washout period.
Groups:
- Zegerid, Prilosec, Sodium Bicarbonate: Participants received Zegerid Oral Suspension (omeprazole 20 mg and sodium bicarbonate 1680 mg) in the first intervention, Prilosec over-the-counter (OTC) Tablets (omeprazole 20 mg) in the second intervention (after washout period), and Sodium Bicarbonate Oral Suspension (sodium bicarbonate 1680 mg) in the third intervention (after washout period)
- Prilosec, Zegerid, Sodium Bicarbonate: Participants received Prilosec OTC Tablets (omeprazole 20 mg) in the first intervention, Zegerid Oral Suspension (omeprazole 20 mg and sodium bicarbonate 1680 mg) in the second intervention (after washout period), and Sodium Bicarbonate Oral Suspension (sodium bicarbonate 1680 mg) in the third intervention (after washout period)
- Zegerid, Prilosec: Participants received Zegerid Oral Suspension (omeprazole 20 mg and sodium bicarbonate 1680 mg) in the first intervention and Prilosec OTC Tablets (omeprazole 20 mg) in the second intervention (after washout period)
- Prilosec, Zegerid: Participants received Prilosec OTC Tablets (omeprazole 20 mg) in the first intervention and Zegerid Oral Suspension (omeprazole 20 mg and sodium bicarbonate 1680 mg) in the second intervention (after washout period)
Period: First Intervention
Arm/Group | Zegerid, Prilosec, Sodium Bicarbonate | Prilosec, Zegerid, Sodium Bicarbonate | Zegerid, Prilosec | Prilosec, Zegerid
Started | 14 | 16 | 14 | 16
Completed | 14 | 16 | 14 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | Zegerid, Prilosec, Sodium Bicarbonate | Prilosec, Zegerid, Sodium Bicarbonate | Zegerid, Prilosec | Prilosec, Zegerid
Started | 14 | 16 | 14 | 16
Completed | 14 | 16 | 14 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Zegerid, Prilosec, Sodium Bicarbonate | Prilosec, Zegerid, Sodium Bicarbonate | Zegerid, Prilosec | Prilosec, Zegerid
Started | 14 | 16 | 14 | 16
Completed | 14 | 16 | 14 | 16
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period of 2 Weeks
Arm/Group | Zegerid, Prilosec, Sodium Bicarbonate | Prilosec, Zegerid, Sodium Bicarbonate | Zegerid, Prilosec | Prilosec, Zegerid
Started | 14 | 16 | 0 | 0
Completed | 14 | 16 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention
Arm/Group | Zegerid, Prilosec, Sodium Bicarbonate | Prilosec, Zegerid, Sodium Bicarbonate | Zegerid, Prilosec | Prilosec, Zegerid
Started | 14 | 16 | 0 | 0
Completed | 14 | 16 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (4.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Median 24-hour Intragastric pH on the 7th Day of Drug Administration
Description: The change from Baseline in median pH was calculated as: median pH on Day 7 minus median pH at Baseline. PH measures how acidic or basic a substance is. The pH scale ranges from 0 to 14. A pH of 7 is neutral. A pH less than 7 is acidic. A pH greater than 7 is basic.
Time Frame: Baseline and 7 days
Population: 25 participants in each arm had good quality tracings and were included in the efficacy analysis.
Measure: Median (Full Range); unit: pH scale
Groups:
- Zegerid: Participants in the 7-Day Dosing group. Measurements taken on the 7th day of Zegerid administration.
- Prilosec: Participants in the 7-Day Dosing group. Measurements taken on the 7th day of Prilosec administration.
Arm/Group | Zegerid | Prilosec
Number analyzed (Participants) | 25 | 25
pH scale
  Day 7 Score | 3.250 (1.300) [1.23 to 5.30] | 4.160 (1.260) [1.46 to 5.78]
  Change from Baseline in PH | 2.180 (1.320) [-0.13 to 4.30] | 2.900 (1.244) [0.10 to 4.21]

ADVERSE EVENTS:
Groups:
- Sodium Bicarbonate (1-Day Dosing): Following completion of the 1-day dosing 2-way crossover study, and a subsequent washout period (minimum of 2 weeks), all participants then received a single administration of sodium bicarbonate 1680 mg.
Arm/Group | Zegerid (7-Day Dosing) | Prilosec (7-Day Dosing) | Sodium Bicarbonate (1-Day Dosing) | Zegerid (1-Day Dosing) | Prilosec (1-Day Dosing)
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 2/30 | 0/30 | 0/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zegerid (7-Day Dosing) (N=30) | Prilosec (7-Day Dosing) (N=30) | Sodium Bicarbonate (1-Day Dosing) (N=30) | Zegerid (1-Day Dosing) (N=30) | Prilosec (1-Day Dosing) (N=30)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other